CLINICAL TRIAL: NCT01042171
Title: Evaluation of Image Quality Over Time After Injection of the ﬂuorescein Sodium for Confocal Laser Endomicroscopy
Status: Completed | Type: Observational
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Chief of the Department of Gastroenterology, Qilu Hospital, Shandong University
Other Study IDs: 2009SDU-QILU-G07
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Change of Image Quality of CLE

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Confocal laser endomicroscopy (CLE) is a newly developed endoscopic technique. The most commonly used fluorescent substance is Fluorescein sodium.The plasma half-life of ﬂuorescein is 11 minutes. A recent test estimated that ﬂuorescein-based CLSM(confocal laser scanning microscopy) of the upper-GI tract of pigs delivers the best contrast and image quality within the ﬁrst 8 minutes after injection of ﬂuorescein .However, despite its increasing use in clinical examination,there are no data on contrast dynamics and image quality over time after injection of the ﬂuorescein sodium in the inspection of gastrointestinal tract of human being.

ELIGIBILITY:
Inclusion Criteria:

* These subjects will include male or female aged between 18 and 60 years with indications for upper-endoscopy ,but without serious gastritis and other serious stomach lesions

Exclusion Criteria:

* Complications such as gastric and/or duodenal peptic ulcer, stenosis
* Esophageal, gastric or duodenal cancer or other malignancy
* History of stomach surgery
* A history of bronchial asthma, or known allergy to fluorescein.
* Pregnant or breast-feeding (for females)
* Below 18 or above 60 years of age
* Severe comorbidities ( e.g. such as renal failure, congestive cardiac failure, liver cirrhosis).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: patients without any disease of heart,liver or kidney;patients without serious gastritis and other serious stomach lesions.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-12; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The ideal time period for the best CLE imaging when using ﬂuorescein sodium is about 10 minutes | Within the 30 minutes after injection of fluorescein

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, PhD. MD., Study Director — Department of Gastroenterology, Qilu Hospital
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China